CLINICAL TRIAL: NCT04382651
Title: A Phase 2, Randomized, Placebo-controlled, Participant and Investigator Blinded, Multi-center Study to Assess Efficacy and Safety of MAS825 for the Treatment of SARS-CoV-2 Infected Patients With COVID-19 Pneumonia and Impaired Respiratory Function
Brief Title: Study of Efficacy and Safety of MAS825 in Patients With COVID-19
Acronym: MAS-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMAS825F12201
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: COVID-19 Pneumonia, Impaired Respiratory Function
Keywords: COVID-19; pneumonia; SARS-Cov2; APACHE II; MAS825; inflammasome
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19; Pneumonia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAS825 + SoC (Experimental): Single dose of MAS825 10 mg/kg by intravenous infusion in addition to SoC
  Interventions: Drug: MAS825; Drug: Standard of Care (SoC)
- Placebo + SoC (Placebo Comparator): Single dose of matching Placebo by intravenous infusion in addition to SoC
  Interventions: Other: Placebo; Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: MAS825 — MAS825 liquid solution for intravenous infusion
  Arms: MAS825 + SoC
Other: Placebo — Placebo liquid solution for intravenous infusion
  Arms: Placebo + SoC
Drug: Standard of Care (SoC) — SoC included a variety of supportive therapies that ranged from the administration of supplementary oxygen to full intensive care support, alongside the use of antiviral treatment, convalescent plasma, corticosteroids, antibiotics or other agents.

SUMMARY:
This clinical study was designed to assess the efficacy and safety of MAS825 for the treatment of severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2) infected patients with coronavirus disease 2019 (COVID-19) pneumonia and impaired respiratory function.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, placebo -controlled, participant and investigator blinded, multi-center study to assess efficacy and safety of MAS825 for the treatment of SARS-CoV-2 infected patients with COVID-19 pneumonia and impaired respiratory function.

The study consisted of five study periods:

Screening / Baseline / Treatment visit (Day -1 to 1): Lasted up to a maximum of 24 hours and comprised a screening / baseline assessment. This visit was used to confirm that the study inclusion and exclusion criteria were met and served as baseline assessment prior to randomization. Participants were randomized as soon as possible, but within a maximum of 24 hours after screening in a 1:1 ratio receiving a single intravenous infusion of MAS825 or placebo in addition to standard of care (SoC) on Day -1 to 1.

Treatment period (Day 2-15): Study assessments were conducted every 2 days for hospitalized participants. If participants were discharged from the hospital prior to Day 15, assessments on the day of discharge were performed according to the schedule listed under Day 15 and those participants returned to the site for the Day 15 assessment (all other visits between discharge and Day 15 were omitted).

Follow-up (Day 16-29): After completion of the treatment period, participants were observed until Day 29 or discharged from hospital, whichever was sooner. Study assessments were conducted every 2 days for domiciled participants. If participants were discharged from hospital prior to Day 29, a study visit conducted by telephone was performed on Day 29 (all other visits between discharge and Day 29 were omitted).

Safety follow-up visit assessment (Day 45): A follow-up visit for safety was conducted at Day 45 if the participant was hospitalized. If participants were discharged from the hospital prior to Day 45, a study visit was conducted by telephone on Day 45.

End of Study/Safety follow-up visit assessment (Day 127): A follow-up visit for safety was conducted at Day 127 if the participant was hospitalized. If participants were discharged from the hospital prior to Day 127, a study visit was conducted by telephone on Day 127.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥18 years at screening
2. Signed Informed Consent Form (ICF) by patient capable of giving consent, or, when the patient is not capable of giving consent, by his or her legal/authorized representative (if allowed according to local requirements)
3. Clinically diagnosed with the SARS-CoV-2 virus by polymerase chain reaction (PCR) or by other approved diagnostic methodology within 7 days prior to randomization
4. Hospitalized with COVID-19-induced pneumonia evidenced by chest x-ray, computed tomography scan (CT scan) or magnetic resonance scan (MR scan) (taken within 5 days prior to randomization)
5. Impaired respiratory function, defined as peripheral oxygen saturation (SpO2) ≤93% on room air or partial pressure of oxygen (PaO2) / fraction of inspired oxygen (FiO2) <300 millimeter of mercury (mmHg) at time of screening For cities located at altitudes greater than 2500 m above sea level, these will be substituted with SpO2 <90% and PaO2/FiO2 <250 mmHg
6. Acute Physiologic Assessment and Chronic Health Evaluation (APACHE) II score of ≥10 at time of screening
7. CRP ≥20 mg/L or ferritin level ≥600 μg/L at screening
8. Body weight between 45 kg and 145 kg, inclusive, at screening
9. Ability to comply with the study protocol, in the investigator's judgment

Exclusion Criteria:

1. History of hypersensitivity to the investigational treatment or their excipients or to drugs of similar chemical classes
2. Suspected active or chronic bacterial (including Mycobacterium tuberculosis), fungal, viral, or other infection with the exception of SARS-CoV-2
3. In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatment
4. Intubated prior to randomization
5. Patients who have explicitly expressed the wish not to receive intensive care support when this would be indicated based on their condition
6. Previous treatment with anti-rejection and immunomodulatory drugs within the past 2 weeks, or within the past 30 days or 5 half-lives (whichever is the longer) for immunomodulatory therapeutic antibodies or prohibited drugs, with the exception of anti-viral therapies or corticosteroids

   * For COVID-19 infection, ongoing corticosteroid treatment is permitted at doses as per local SoC
   * For non-COVID-19 disorders, ongoing corticosteroid treatment is permitted at doses up to and including prednisolone 10 mg daily or equivalent.
7. Serum alanine transaminase (ALT) or aspartate transaminase (AST) >5 times upper limit of normal detected within 24 hours at screening/baseline (according to local laboratory reference ranges) or other evidence of severe hepatic impairment.
8. Absolute peripheral blood neutrophil count of ≤1000/mm^3
9. Estimated GFR (eGFR) ≤30 mL/min/1.73m^2 (based on CKD-EPI formula)
10. Pregnant or breastfeeding, or positive urine or serum pregnancy test in a pre-dose examination
11. Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they agree to abstain from any sexual intercourse for a total of 29 days after randomization (the 14-day treatment period plus a 14-day follow-up period).
13. Current participation in any other investigational trials, with the exception of (not yet) approved COVID-19 therapies that are considered (local) standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- United States (20):
  - Novartis Investigative Site, Chula Vista, California
  - Novartis Investigative Site, Glendale, California
  - Novartis Investigative Site, Irvine, California
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Idaho Falls, Idaho
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Brooklyn, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Bend, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Mesquite, Texas

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Hakim AD, Awili M, O'Neal HR, Siddiqi O, Jaffrani N, Lee R, Overcash JS, Chauffe A, Hammond TC, Patel B, Waters M, Criner GJ, Pachori A, Junge G, Levitch R, Watts J, Koo P, Sengupta T, Yu L, Kiffe M, Pinck A, Stein RR, Bendrick-Peart J, Jenkins J, Rowlands M, Waldron-Lynch F, Matthews J. Efficacy and safety of MAS825 (anti-IL-1beta/IL-18) in COVID-19 patients with pneumonia and impaired respiratory function. Clin Exp Immunol. 2023 Oct 13;213(3):265-275. doi: 10.1093/cei/uxad065. PMID 37338154
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 21 investigative sites in 1 country, United States.
Pre-assignment Details: The participants were screened within 24 hours prior to enrollment. The single dose was administered within a maximum of 24 hours after screening and baseline assessments.
Period: Overall Study
Arm/Group | MAS825 + SoC | Placebo + SoC
Started (All randomized participants) | 69 | 71
Safety Analysis Set (All randomized participants that have received any study drug) | 68 | 70
Pharmacokinetics (PK) Analysis Set (All randomized participants with at least one valid PK concentration measurement, who received MAS825 and no protocol deviations with relevant impact on PK data.) | 63 | 0
Completed | 38 | 43
Not Completed | 31 | 28
Not completed — Death | 26 | 23
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MAS825 + SoC | Placebo + SoC | Total
Number analyzed (Participants) | 69 | 71 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (12.46) | 63.7 (12.91) | 64.5 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 39 | 48 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 6 | 8 | 14
  White | 51 | 52 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: APACHE II Severity of Disease Score on Day 15 or on the Day of Discharge (Whichever is Earlier)
Description: The APACHE II ("Acute Physiology And Chronic Health Evaluation II") is a severity-of-disease classification system. An integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death. In practice, it is rare for any participant to accumulate more than 55 points.
  APACHE II score was measured on Day 15 or on the day of discharge (whichever was earlier). Participants who died on Day 15 or earlier were assigned the highest observed APACHE II score of any of the participants at any time during the trial (worst case imputation for deaths). Missing data values of the parameters required for the derivation of the APACHE II score were replaced by the last available assessment.
Time Frame: up to Day 15
Population: Safety Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | MAS825 + SoC | Placebo + SoC
Number analyzed (Participants) | 68 | 70
Score on a scale | 14.5 (1.87) | 13.5 (1.8)
Statistical Analysis 1: Comparison: MAS825 + SoC vs Placebo + SoC; Test type: Superiority; p = 0.33, ANCOVA — 1-Sided; Mean Difference (Final Values) = 0.98, 90% CI 2-sided [-2.7 to 4.7], Standard Error of Mean 2.225

2. Secondary Outcome: Serum C-reactive Protein (CRP) Levels
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. It was analyzed on a log-scale fitting a repeated measures mixed model: treatment, visit, stratification factors, visit * treatment and visit * stratification factors as fixed effects and log-transformed baseline score and visit * log-transformed baseline score as continuous covariate. Values reported were back-transformed to original scale.
Time Frame: Baseline, days 2, 4, 6, 8, 10, 12, 14 and 15
Population: Safety Analysis Set
Measure: Geometric Least Squares Mean (Standard Error); unit: Milligram / Liter
Arm/Group | MAS825 + SoC | Placebo + SoC
Number analyzed (Participants) | 68 | 70
Milligram / Liter
  Day 2: number analyzed (Participants) | 61 | 67
  Day 2 | 55.50 (1.11) | 57.70 (1.10)
  Day 4: number analyzed (Participants) | 55 | 58
  Day 4 | 28.30 (1.19) | 37.10 (1.19)
  Day 6: number analyzed (Participants) | 53 | 47
  Day 6 | 19.80 (1.24) | 22.30 (1.24)
  Day 8: number analyzed (Participants) | 40 | 42
  Day 8 | 15.00 (1.31) | 16.6 (1.30)
  Day 10: number analyzed (Participants) | 37 | 39
  Day 10 | 10.10 (1.38) | 19.80 (1.35)
  Day 12: number analyzed (Participants) | 29 | 30
  Day 12 | 11.00 (1.42) | 15.80 (1.39)
  Day 14: number analyzed (Participants) | 25 | 24
  Day 14 | 7.30 (1.43) | 13.20 (1.39)
  Day 15: number analyzed (Participants) | 39 | 42
  Day 15 | 5.70 (1.40) | 11.60 (1.36)

3. Secondary Outcome: Ferritin Levels
Description: Ferritin is a blood test marker for inflammation in the body. For a standard ferritin test, a normal reading is less than 300 micrograms per liter (μg/L). It was analyzed on a log-scale fitting a repeated measures mixed model: treatment, visit, stratification factors, visit * treatment and visit * stratification factors as fixed effects and log-transformed baseline score and visit * log-transformed baseline score as continuous covariate. Values reported were back-transformed to original scale.
Time Frame: Baseline, days 2, 4, 6, 8, 10, 12, 14 and 15
Population: Safety Analysis Set
Measure: Geometric Least Squares Mean (Standard Error); unit: Microgram / Liter
Arm/Group | MAS825 + SoC | Placebo + SoC
Number analyzed (Participants) | 68 | 70
Microgram / Liter
  Day 2: number analyzed (Participants) | 65 | 68
  Day 2 | 773.20 (1.05) | 800.20 (1.05)
  Day 4: number analyzed (Participants) | 57 | 58
  Day 4 | 692.70 (1.05) | 701.40 (1.05)
  Day 6: number analyzed (Participants) | 52 | 47
  Day 6 | 687.50 (1.10) | 622.10 (1.10)
  Day 8: number analyzed (Participants) | 42 | 42
  Day 8 | 674.00 (1.12) | 667.80 (1.11)
  Day 10: number analyzed (Participants) | 36 | 39
  Day 10 | 670.00 (1.16) | 776.00 (1.15)
  Day 12: number analyzed (Participants) | 30 | 30
  Day 12 | 680.00 (1.18) | 754.50 (1.17)
  Day 14: number analyzed (Participants) | 25 | 24
  Day 14 | 541.70 (1.22) | 595.70 (1.22)
  Day 15: number analyzed (Participants) | 34 | 34
  Day 15 | 502.90 (1.21) | 504.20 (1.21)

4. Secondary Outcome: Number of Participants Not Requiring Mechanical Ventilation for Survival
Description: Number of participants not requiring mechanical ventilation for survival until Day 15 and Day 29: defined by WHO 9-point ordinal scale score of < 6 points at all time points assessments.
  The scoring is - Uninfected patients have a score 0. - Ambulatory patients can have a score 1 (no limitation of activities) or 2 (limitation of activities). - Hospitalized patients with mild disease can have score 3 (no oxygen therapy) or 4 (oxygen by mask or nasal prongs). - Hospitalized patients with severe disease can have score 5 (non-invasive ventilation or high-flow oxygen), 6 (intubation and mechanical ventilation) or 7 (ventilation + additional organ support). - Patients who die have a score 8.
  Missing data values were handled as follows: For participants who died prior to Day 29, the score for death was imputed for all following visits up to and including Day 29. For all the other participants, last observation carried forward was applied up to and including Day 29.
Time Frame: Until Day 15 (Assessments on Days 2, 4, 6, 8, 10, 12, 14 and 15) and until Day 29 (Additional assessments on Days 17, 19, 21, 23, 25, 27 and 29)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MAS825 + SoC | Placebo + SoC
Number analyzed (Participants) | 68 | 70
Participants
  Until Day 15 | 41 | 47
  Until Day 29 | 39 | 45

5. Secondary Outcome: Number of Participants With at Least One-point Improvement From Baseline in Clinical Status
Description: Number of participants with at least one-point improvement from baseline in clinical status, which was measured with WHO 9-point ordinal scale.
  The scoring is - Uninfected patients have a score 0. - Ambulatory patients can have a score 1 (no limitation of activities) or 2 (limitation of activities). - Hospitalized patients with mild disease can have score 3 (no oxygen therapy) or 4 (oxygen by mask or nasal prongs). - Hospitalized patients with severe disease can have score 5 (non-invasive ventilation or high-flow oxygen), 6 (intubation and mechanical ventilation) or 7 (ventilation + additional organ support). - Patients who die have a score 8.
  Missing data values were handled as follows: For participants who died prior to Day 29, the score for death was imputed for all following visits up to and including Day 29. For all the other participants, last observation carried forward was applied up to and including Day 29.
Time Frame: Baseline, Day 15 and Day 29
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MAS825 + SoC | Placebo + SoC
Number analyzed (Participants) | 68 | 70
Participants
  Day 15 | 39 | 39
  Day 29 | 43 | 46

6. Secondary Outcome: Clinical Status Over Time
Description: Clinical status was measured with World Health Organization (WHO) 9-point ordinal scale.
  The scoring is - Uninfected patients have a score 0. - Ambulatory patients can have a score 1 (no limitation of activities) or 2 (limitation of activities). - Hospitalized patients with mild disease can have score 3 (no oxygen therapy) or 4 (oxygen by mask or nasal prongs). - Hospitalized patients with severe disease can have score 5 (non-invasive ventilation or high-flow oxygen), 6 (intubation and mechanical ventilation) or 7 (ventilation + additional organ support - pressors, renal replacement therapy, extracorporeal membrane oxygenation). - Patients who die have a score 8.
  Missing data values were handled as follows: For participants who died prior to Day 127, the score for death was imputed for all following visits up to and including Day 127. For all the other participants, last observation carried forward was applied up to and including Day 127.
Time Frame: Baseline, days 2, 4, 6, 8, 10, 12, 14, 15, 17, 19, 21, 23, 25, 27, 29, 45 and 127
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MAS825 + SoC | Placebo + SoC
Number analyzed (Participants) | 68 | 70
Score on a scale
  Baseline | 4.8 (0.38) | 4.7 (0.49)
  Day 2 | 4.8 (0.71) | 4.7 (0.57)
  Day 4 | 4.8 (0.90) | 4.7 (1.13)
  Day 6 | 4.8 (1.27) | 4.7 (1.40)
  Day 8 | 4.9 (1.63) | 4.5 (1.64)
  Day 10 | 4.9 (1.76) | 4.6 (1.80)
  Day 12 | 5.0 (1.97) | 4.7 (2.04)
  Day 14 | 5.0 (2.04) | 4.8 (2.09)
  Day 15 | 4.5 (2.59) | 4.2 (2.58)
  Day 17 | 4.4 (2.64) | 4.2 (2.67)
  Day 19 | 4.4 (2.73) | 4.1 (2.70)
  Day 21 | 4.4 (2.78) | 4.1 (2.71)
  Day 23 | 4.4 (2.78) | 4.1 (2.73)
  Day 25 | 4.4 (2.79) | 4.2 (2.76)
  Day 27 | 4.4 (2.81) | 4.2 (2.76)
  Day 29 | 4.2 (2.99) | 3.8 (3.00)
  Day 45 | 4.0 (3.19) | 3.7 (3.24)
  Day 127 | 3.8 (3.48) | 3.3 (3.41)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of administration of study treatment to day 127.
Description: Any sign or symptom that occurs during the study treatment plus the 127 days post treatment.
Groups:
- Total: Total
Arm/Group | MAS825 + SoC | Placebo + SoC | Total
All-Cause Mortality (participants affected / at risk) | 26/68 | 23/70 | 49/138
Serious Adverse Events (participants affected / at risk) | 31/68 | 28/70 | 59/138
Other Adverse Events (participants affected / at risk) | 20/68 | 19/70 | 39/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAS825 + SoC (N=68) | Placebo + SoC (N=70) | Total (N=138)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 2
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 2 | 3 | 5
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 1 | 2
Myocarditis (Cardiac disorders) | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Hypothermia (General disorders) | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 2 | 1 | 3
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 2 | 4 | 6
Fungaemia (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 2 | 1 | 3
Septic shock (Infections and infestations) | 3 | 0 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 3
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 4 | 7
Nephropathy (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 6
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 8 | 19
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 6
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 10
Distributive shock (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 1 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MAS825 + SoC (N=68) | Placebo + SoC (N=70) | Total (N=138)
Atrial fibrillation (Cardiac disorders) | 4 | 4 | 8
Pneumonia bacterial (Infections and infestations) | 6 | 2 | 8
Urinary tract infection (Infections and infestations) | 2 | 5 | 7
Transaminases increased (Investigations) | 0 | 5 | 5
Anxiety (Psychiatric disorders) | 3 | 6 | 9
Acute kidney injury (Renal and urinary disorders) | 9 | 5 | 14
Hypotension (Vascular disorders) | 5 | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT04382651/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT04382651/SAP_001.pdf